CLINICAL TRIAL: NCT02047344
Title: A Single-Arm, Open-Label, Phase II Trial Evaluating the Efficacy, Safety and Pharmacokinetics of Antroquinonol in Patients With Stage IV (Including Pleural Effusion) Non Squamous NSCLC Who Have Failed Two Lines of Anti-Cancer Therapy
Brief Title: Efficacy, Safety and Pharmacokinetics Study of Antroquinonol to Treat NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Golden Biotechnology Corporation (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHNSCLC-2 001
Record Dates: First submitted 2014-01-16; First posted 2014-01-28 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Non-small Cell Lung Cancer Stage IV
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — antroquinonol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antroquinonol (Hocena) (Experimental): patients will receive one 12 week cycle of antroquinonol 200 mg t.i.d. or until disease progression, unacceptable toxicity, non compliance or withdrawal of consent by the patient, or the investigator decides to discontinue treatment, whichever comes first.
  Interventions: Drug: Antroquinonol

INTERVENTIONS:
Drug: Antroquinonol — patients will receive one 12 week cycle of antroquinonol 200 mg t.i.d. or until disease progression, unacceptable toxicity, non compliance or withdrawal of consent by the patient, or the investigator decides to discontinue treatment, whichever comes first.
  Other Names: Hocena

SUMMARY:
This is a single arm, open label, Phase II study in KRAS-positive and KRAS-negative patients with stage IV (including pleural effusion) non squamous NSCLC who have failed two lines of anti-cancer therapy. A maximum of 60 evaluable patients with NSCLC will receive antroquinonol, of which 30 patients will be KRAS-positive and 30 patients KRAS-negative. An evaluable patient will have received at least one dose of antroquinonol and have a valid baseline tumor assessment. Enrollment will continue until the target number of evaluable patients has been enrolled.

DETAILED DESCRIPTION:
1. Progression free survival rate at 12 weeks, defined as the proportion of patients alive and progression free at Week 12. Patients will be progression free if they have no tumor assessments of progressive disease (defined according to RECIST guidelines, version 1.1) at any point from the start of treatment to Week 12.
2. Objective response rate (ORR), defined as the proportion of patients whose best overall response is either CR or PR according to RECIST version 1.1. The best overall response is the best response recorded during the first 12 week treatment cycle.
3. Disease control rate (DCR), defined as the proportion of patients with a documented CR, PR and SD during the first 12 week treatment cycle according to RECIST version 1.1.
4. Duration of overall tumor response (DR), defined as the interval between the date of the first observation of tumor response (CR or PR) and the date of disease progression or death.
5. Progression free survival defined as the time from randomization to objective tumor progression by RECIST version 1.1 or death due to any cause, whichever occurs first.
6. Overall survival (OS) defined as the time from randomization to death from any cause.
7. Time to progression (TTP) defined as the time from randomization to objective tumor progression by RECIST version 1.1.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed non squamous NSCLC Stage IV (including pleural effusion).
* Radiologically confirmed disease progression following two previous lines of anti-cancer therapy, one of which should be a platinum based regimen, OR the patient has refused treatment with approved treatment modalities
* At least one radiologically measurable target lesion per RECIST version 1.1
* Fresh or archival biopsy tissue available to determine tumor mutation status
* Written informed consent that is consistent with International Conference on Harmonisation Tripartite Guideline on Good Clinical Practice guidelines
* Patient or legally acceptable representative has granted written informed consent before any study specific procedures (including special Screening tests) are performed
* Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1 or 2
* Hemoglobin ≥ 9.0 g/dL; platelets ≥ 100 x 109/L; absolute neutrophil count ≥ 1.5 x 109/L without the use of hematopoietic growth factors
* Bilirubin and creatinine less than 2 × upper limit of normal (ULN) for the institution
* Albumin ≥ 2.5 mg/dL
* Aspartate aminotransferase and alanine aminotransferase less than 5 × ULN for the institution
* Prothrombin time less than 1.5 × ULN for the institution
* Potassium, magnesium and phosphorus within the normal range for the institution (supplementation is permissible)
* Recovery to Grade 1 or baseline of any toxicities due to prior treatments, excluding alopecia

Exclusion Criteria:

* Chemo-, hormone- or immunotherapy, within 4 weeks or within less than four half lives of the date of first administration of study drug and/or persistence of toxicities of prior anti-cancer therapies which are deemed to be clinically relevant
* Radiotherapy within the past 2 weeks prior to date of first administration of study drug
* Previous treatment with an histone deacetylase inhibitor or an epidermal growth factor receptor inhibitor within at least 4 weeks of the date of first administration of study drug
* Treatment with any drug(s) known to be an inhibitor or inducer of cytochrome P450 (CYP)2C19, CYP3A4, CYP2C8, and CYP2E1, within 14 days of the date of first administration of study drug
* Brain metastases, which are symptomatic; patients with treated, brain metastases are eligible with stable brain disease for at least 4 weeks without the requirement for steroids or anti epileptic therapy
* Inability to swallow oral medications or a recent acute gastrointestinal disorder with diarrhea e.g., Cohn's disease, malabsorption, or Common Terminology Criteria for Adverse Event (CTCAE) Grade > 2 diarrhea of any etiology at baseline
* Other malignancies diagnosed within the past five years (other than curatively treated cervical cancer in situ), non melanoma skin cancer, superficial bladder tumors Ta (non invasive tumor) and TIS (carcinoma in situ)
* Patients with any serious active infection (i.e., requiring an intravenous antibiotic, antifungal, or antiviral agent)
* Patients with known human immunodeficiency virus, active hepatitis B or active hepatitis C
* Patients who have any other life threatening illness or organ system dysfunction, which in the opinion of the investigator, would either compromise patient safety or interfere with the evaluation of the safety of the study drug
* Known or suspected substance abuse or alcohol abuse
* Pregnancy or breast feeding
* History of clinically significant or uncontrolled cardiac disease, including congestive heart failure, angina, myocardial infarction, arrhythmia, including New York Heart Association functional classification of three

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-10; Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Cheng, Ph.D., Study Director — Golden Biotechnology Corp.
Locations (10):
- United States (7):
  - Arizona Clinical Research Center, Tucson, Arizona
  - UCSF, San Francisco, California
  - Rush University Medical Center, Chicago, Illinois
  - John Hopkins University, Baltimore, Maryland
  - Peninsula Regional Med Center, Salisbury, Maryland
  - Henry Ford health system, Detroit, Michigan
  - Guthrie Clinic, Ltd, Sayre, Pennsylvania
- Taiwan (3):
  - Chang Gung Memorial Hospital-Kaohsiung medical center, Kaohsiung City
  - National Cheng Kung University Hospitail, Tainan
  - Tri Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
need DMC proved

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Unselected KRAS-positive and KRAS-negative patients with stage IV (including pleural effusion) non squamous NSCLC and radiologically-confirmed disease progression following greater than or equal to two, but less than or equal to four, prior lines of systemic anti cancer therapy.
Pre-assignment Details: Written informed consent was obtained from all patients before initiating screening. The screening period was up to 42 days in duration (Days 42 to 1) for K-Ras testing result, if no history k-Ras result.
Groups:
- K-Ras Negative: Fresh or archival biopsy tissue to determine KRAS is not mutant.
- K- Ras Mutant: Fresh or archival biopsy tissue to determine KRAS is mutant.
Period: Overall Study
Arm/Group | K-Ras Negative | K- Ras Mutant
Started | 16 (one patient is not evaluable in process. however, evaluable to safety report.) | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- K-Ras Negative: Fresh or archival biopsy tissue to determine KRAS is not mutant. Patients will receive one 12 week cycle of antroquinonol 200 mg t.i.d. or until disease progression.
- K- Ras Mutant: Fresh or archival biopsy tissue to determine KRAS is mutant. Patients will receive one 12 week cycle of antroquinonol 200 mg t.i.d. or until disease progression.
- Total: Total of all reporting groups
Arm/Group | K-Ras Negative | K- Ras Mutant | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 9 | 12 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 11 | 8 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 1 | 9
  Black or African American | 1 | 1 | 2
  White | 6 | 13 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 14 | 21
  Taiwan | 8 | 1 | 9
ECOG performance status [Count of Participants; unit: Participants]
  Fully active | 10 | 1 | 11
  Restricted in physically strenuous activity | 4 | 12 | 16
  Capable of all selfcare more than 50% work | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate
Description: Tumor response will be assessed at 6 week intervals during the first treatment cycle using the RECIST criteria, version 1.1. Each patient will be assigned one of the following categories: 1) complete response (CR), 2) partial response (PR), 3) stable disease (SD), or 4) progressive disease (PD). Patients who died from any cause or discontinued the study for any reason without a post screening or Week 12 tumor assessment will be considered as failing to respond to treatment.
Time Frame: 12 weeks
Population: Defined as the proportion of patients alive and progression free at Week 12.
Measure: Count of Participants; unit: Participants
Groups:
- Progression-free Survival Rate/KRAS Negative Group; Progression-free Survival Rate/KRAS Mutant Group: 200mg TID for treating KRAS negative patients 12 weeks
Arm/Group | Progression-free Survival Rate/KRAS Negative Group | Progression-free Survival Rate/KRAS Mutant Group
Number analyzed (Participants) | 15 | 15
Participants | 4 | 0

2. Secondary Outcome: Cmax
Description: PK sampling will be performed on Days 0 and 28 in all patients enrolled in Stage 1.PK endpoints will be derived for intensively sampled PK profiles by non compartmental methods and include: Cmax: peak concentration;Ctrough: trough plasma concentration.
Time Frame: 8 hours
Population: There were 22 patients with reported concentration data who were eligible for the PK population.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Antroquinonol Day 28: continue use Antroquinonol for 28 Days
Arm/Group | Antroquinonol (Hocena) | Antroquinonol Day 28
Number analyzed (Participants) | 22 | 22
ng/mL | 276.87 (211.162) | 393.55 (315.434)

3. Secondary Outcome: Disease Control Rate (DCR)
Description: the proportion of patients with a documented CR, PR and SD during the first 12 week treatment cycle according to RECIST version 1.1.
Time Frame: 12 weeks
Population: 26 patients can be run the full analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Non- Prior Chemotherapies: Patient without any chemotherapy before join Study
- One Line Failed Prior Chemotherapies: Patient join with One line failed prior chemotherapies
- Two Lines Failed Prior Chemotherapies: Patients join with two lines failed prior chemotherapies
- More Than Two Lines Failed Prior Chemotherapies: patient failed more than two line chemotherapies before join.
Arm/Group | Non- Prior Chemotherapies | One Line Failed Prior Chemotherapies | Two Lines Failed Prior Chemotherapies | More Than Two Lines Failed Prior Chemotherapies
Number analyzed (Participants) | 5 | 3 | 7 | 11
percentage of participants | 40 [5.3 to 85.3] | 0 [0 to 70.8] | 42.9 [9.9 to 81.6] | 72.7 [39.0 to 94.0]

4. Secondary Outcome: T½: the Time Required for a Quantity to Reduce to Half Its Initial Value
Description: PK sampling will be performed on Days 0 and 28 in all patients enrolled in Stage 1.PK endpoints will be derived for intensively sampled PK profiles by T½: terminal half life
Time Frame: 8 hours
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | Antroquinonol (Hocena) | Antroquinonol Day 28
Number analyzed (Participants) | 22 | 22
hours | 3 [0.5 to 4] | 2 [0.5 to 4]

5. Other Pre Specified Outcome: Objective Response Rate (ORR)
Description: Defined as the proportion of patients whose best overall response is either CR or PR according to RECIST version 1.1. The best overall response is the best response recorded during the first 12 week treatment cycle.
Time Frame: 12 weeks
Population: full sey analysis group
Measure: Number; unit: patients
Arm/Group | Antroquinonol (Hocena)
Number analyzed (Participants) | 26
patients | 0

6. Other Pre Specified Outcome: Overall Survival
Description: the time from the date of first administration of study drug to death from any cause
Time Frame: up to week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non- Prior Chemotherapies | One Line Failed Prior Chemotherapies | Two Lines Failed Prior Chemotherapies | More Than Two Lines Failed Prior Chemotherapies
Number analyzed (Participants) | 5 | 3 | 7 | 11
percentage of participants
  week 12 | 60 [12.6 to 88.2] | 100 [100 to 100] | 100 [100 to 100] | 90.9 [50.8 to 98.7]
  week 48 | 0 [0 to 0] | 100 [100 to 100] | 28.6 [4.1 to 61.2] | 39.3 [7.3 to 71.6]

ADVERSE EVENTS:
Time Frame: AEs collected for up to 48 weeks of the study from the time the patient signed the informed consent.
Description: Patients were followed for AEs from the date of informed consent until resolution or stabilization, alternative treatment for NSCLC was started 6 months after last dose of study drug, or loss to follow-up, whichever occurred first. In the event of serious or study drug-related toxicities, the patient was followed until resolution or stabilization. Safety follow up data was collected by telephone contact every 3 months after the EOS visit.
Arm/Group | Antroquinonol (Hocena)
All-Cause Mortality (participants affected / at risk) | 14/31
Serious Adverse Events (participants affected / at risk) | 12/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antroquinonol (Hocena) (N=31)
Cardiac disorders (Cardiac disorders) | 2 (3) — Atrial fibrillation Cardiac arrest Tachycardia
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) — Diarrhoea Intestinal obstruction
General disorders and administration site conditions (General disorders) | 2 (2) — Death Disease progression
Infections and infestations (Infections and infestations) | 4 (4) — Pneumonia Pyelonephritis acute
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2) — Dehydration Hyponatraemia
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) — Malignant neoplasm progression Metastases to central nervous system
Nervous system disorders (Nervous system disorders) | 1 (1) — Dizziness
Renal and urinary disorders (Renal and urinary disorders) | 2 (4) — Haematuria Hydronephrosis Ureteric stenosis Urinoma
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 (5) — Acute respiratory failure Dyspnoea Pulmonary oedema Respiratory distress
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antroquinonol (Hocena) (N=31)
Tachycardia (Cardiac disorders) | 2 (5)
Gastrointestinal disorders (Gastrointestinal disorders) | 30 (30) — Abdominal pain Abdominal pain upper Diarrhoea Flatulence Nausea Vomiting
General disorders and administration site conditions (General disorders) | 20 (20) — Catheter site pain Chest pain Fatigue Influenza like illness
Infections and infestations (Infections and infestations) | 6 (6) — Pneumonia
Investigations (Investigations) | 6 (6) — Urine analysis abnormal Weight decreased
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 11 (11) — Decreased appetite Dehydration Hypomagnesaemia
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 8 (8) — Musculoskeletal pain Pain in extremity
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) — Malignant neoplasm progression
Nervous system disorders (Nervous system disorders) | 11 (11) — Dizziness Headache Neuropathy peripheral
Psychiatric disorders (Psychiatric disorders) | 4 (4) — Insomnia
Renal and urinary disorders (Renal and urinary disorders) | 4 (4) — Haematuria
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 17 (17) — Acute respiratory failure Cough Dyspnoea Nasal congestion Pleural effusion Pneumothorax

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT02047344/Prot_000.pdf
  • Statistical Analysis Plan (2014-08-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT02047344/SAP_001.pdf